CLINICAL TRIAL: NCT04482491
Title: Histological Prediction and Choice of the Resection Strategy in Front of a Colorectal Lesion > 2 cm: Prospective Comparison of Endoscopic Characterization, Non-targeted and Targeted Biopsies
Status: Completed | Type: Observational
Sponsor: Hôpital Edouard Herriot (Other)
Responsible Party: Principal Investigator, Jean Christophe Saurin, Professor, Hôpital Edouard Herriot
Other Study IDs: Endoscopic Characterization
Record Dates: First submitted 2020-07-18; First posted 2020-07-22 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Endoscopic Submucosal Dissection
MeSH Terms: interventions — Endoscopic Mucosal Resection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Endoscopic Submucosal Dissection — Endoscopic Submucosal Dissection

SUMMARY:
Colorectal cancer has become a public health priority considering its increased prevalence and high mortality rate when diagnosed late. As a consequence, many countries have promoted and uptaken of colorectal cancer screening programs leading to an increasing detection of advanced but also superficial lesions ESGE (European Society of Gastrointestinal Endoscopy) guidelines states that the majority of those colonic and rectal superficial lesions can be removed in a curative way by standard polypectomy and/or by EMR (Endoscopic Mucosal Resection) and that ESD (Endoscopic Submucosal Dissection) can be considered for removal of colonic and rectal lesions with high suspicion of limited submucosal invasion. Histologically, a resection is curative for the patient when the adenocarcinoma is well-differentiated (G1/G2), with a depth of invasion ≤ sm1 (≤ 1 mm submucosal invasion), with no lymphovascular invasion nor budding and with lateral and deep margins free of cancer

ELIGIBILITY:
Inclusion Criteria:

Patients with colorectal lesions> 2 cm because any gastroenterologist must be able to resect 2 cm polyps on their own and therefore should never need to take biopsies to clarify the histology before resection.

Patient consenting after information If the lesion is defined by an endoscopist as CONECCT IIA, simple adenoma, the lesion will be resected by en bloc mucosectomy or piece meal depending on its size (after a biopsy, secondary objective).

If the lesion is defined by an endoscopist as CONECCT IIC, adenoma at risk or superficial cancer (<1000µm depth), the lesion will be resected by R0 en bloc by mucosectomy or dissection if the lesion is greater than 20mm (after a biopsy, secondary objective).

If the lesion is defined by an endoscopist as CONECCT III, deep adenocarcinoma (≥1000µm depth), it will be sampled from the most severe part by biopsy forceps and the patient will be referred to oncology or surgery according to the extension assessment .

Pathology available of endoscopic or surgical resection piece Follow-up at 6 months after treatment for CONECCT IS, IIA, IIC lesions by endoscopic control and III by clinical or imaging control.

.

-

Exclusion Criteria:

Metastatic lesion immediately before colonoscopy Patients under guardianship Age <18 Pregnant woman Contraindication to colonoscopy.

-

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Hgh Risk Colorectal Cancer
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
correlation between the histological prediction according to the CONECCT classification, the directed biopsy, the non-directed biopsy and the final histology of the completely resected part (R0). | 1 Year

CONTACTS AND LOCATIONS:
Locations (1):
- Edouard Herriot Hospital, Lyon, Auvergne-Rhône-Alpes, France

IPD SHARING:
Plan to Share IPD: No